CLINICAL TRIAL: NCT04212052
Title: Split-course Hypofractionated Radiotherapy With Concurrent Chemotherapy in Locally Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO 1052
Record Dates: First submitted 2019-12-24; First posted 2019-12-26 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; Split-course radiotherapy; consolidation immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- split-course radiotherapy (Experimental): The radiotherapy is delivered using simultaneous integrated boost (SIB)-intensity-modulated radiotherapy (IMRT). The dose of 30Gy with a fraction dose of 5Gy was delivered to PTV-GTV as the hypo-RT course. Patients were eligible to receive the hypo-boost when there was no disease progression and no persistent ≥G2 treatment-related toxicities. For patients with persistent ≥G2 toxicities, a re-evaluation was planned every 2 weeks to determine whether they were qualified to receive the hypoboost. All eligible patients underwent a repeat 4DCT simulation scan to reformulate the adaptive radiation therapy plan. The adaptive plan of the hypo-boost was delivered to the residual tumor (PTV-GTV-residual) at a dose of 30Gy in 6 fractions (5 Gy per fraction).
  Patients received a weekly infusion of docetaxel (25 mg/m2) and cisplatin (25 mg/m2) concurrent with hypo-RT and hypo-boost therapy. Intended chemotherapy included 4 cycles throughout the course of treatment.
  Interventions: Radiation: split-course radiotherapy; Drug: concurrent chemotherapy; Drug: consolidation immunotherapy

INTERVENTIONS:
Radiation: split-course radiotherapy — The radiotherapy is delivered using simultaneous integrated boost (SIB)-intensity-modulated radiotherapy (IMRT). The dose of 30Gy with a fraction dose of 5Gy was delivered to PTV-GTV as the hypo-RT course. Patients were eligible to receive the hypo-boost when there was no disease progression and no persistent ≥G2 treatment-related toxicities. For patients with persistent ≥G2 toxicities, a re-evaluation was planned every 2 weeks to determine whether they were qualified to receive the hypoboost. All eligible patients underwent a repeat 4DCT simulation scan to reformulate the adaptive radiation therapy plan. The adaptive plan of the hypo-boost was delivered to the residual tumor (PTV-GTV-residual) at a dose of 30Gy in 6 fractions (5 Gy per fraction).
Drug: concurrent chemotherapy — Patients received a weekly infusion of docetaxel (25 mg/m2) and cisplatin (25 mg/m2) concurrent with hypo-RT and hypo-boost therapy. Intended chemotherapy included 4 cycles throughout the course of treatment.
Drug: consolidation immunotherapy — Patients without disease progression or persistent grade2+ toxicities after thoracic radiotherapy were recommended to receive consolidation immunotherapy

SUMMARY:
This Phase II study is to determine the efficacy of split-course thoracic radiotherapy plus concurrent chemotherapy with or without consolidation immunotherapy for patients with local advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
This Phase II study is to determine the efficacy of split-course thoracic radiotherapy plus concurrent chemotherapy with or without consolidation immunotherapy for local advanced non-small cell lung cancer patients.

Patients were treated with hypo-RT (30Gy in 6 fractions) followed by hypo-boost (30Gy in 6 fractions) combined with concurrent weekly chemotherapy (docetaxel 25 mg/m2 and cisplatin 25 mg/m2). Consolidation immunotherapy were recommended for those without disease progression or persistent grade2+ toxicities following radiotherapy. The primary end point is progression-free survival, which is the time that passes from the first day of radiotherapy to the date at which disease progresses. Progression-free survival will be calculated using the Kaplan-Meier method.Toxicities will be graded according to CTCAE v. 5.0.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer (NSCLC) by bronchoscopy, CT-guided biopsy, and endobronchial ultrasonography
* Unresectable stage III disease based on the seventh edition of the TNM (tumor, node, metastases) staging system proposed by the American Joint Committee on Cancer
* Measurable lesions according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1;
* Charlson Comorbidity Index score ≤4
* Previously treated with chemotherapy or treatment-naive
* No previous chest radiotherapy, immunotherapy or biotherapy
* Hemoglobin≥10 mg/dL, platelet≥100000/μL,absolute neutrophil count ≥1500/μL
* Serum creatinine ≤1.25 times the upper normal limit(UNL), or creatinine clearance≥60 ml/min
* Bilirubin ≤1.5 times UNL, AST（SGOT）≤2.5 times UNL ,ALT（SGPT）≤2.5 times UNL,alkaline phosphatase ≤5 times UNL
* CB6 within normal limits
* patients and their family signed the informed consents

Exclusion Criteria:

* Previous or recent another malignancy, except nonmelanoma skin cancer or cervical cancer in situ
* Contraindication for chemotherapy
* Malignant pleural or pericardial effusion.
* Women in pregnancy, lactation period, or no pregnancy test 14 days before the first dose
* Women who has the probability of pregnancy without contraception
* Tendency of hemorrhage
* In other clinical trials within 30 days
* Addicted in drugs or alcohol, AIDS patients
* Uncontrollable seizure or psychotic patients without self-control ability
* Severe allergy or idiosyncrasy
* Not suitable for this study judged by researchers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 2 year

SECONDARY OUTCOMES:
Overall survival | 2 years
response rate | 2 months
rate of grade 3-4 radiation esophagitis | 1 year
rate of grade 3-4 radiation pneumonitis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Ph.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, China

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Schrum D, Carter D, Kelsey C, et al: Non Small Cell Lung Cancer (ed 9). Philadelphia, PA, Lippincott Williams & Wilkins, 2011, pp 799-847.
- [Background] Dillman RO, Seagren SL, Propert KJ, Guerra J, Eaton WL, Perry MC, Carey RW, Frei EF 3rd, Green MR. A randomized trial of induction chemotherapy plus high-dose radiation versus radiation alone in stage III non-small-cell lung cancer. N Engl J Med. 1990 Oct 4;323(14):940-5. doi: 10.1056/NEJM199010043231403. PMID 2169587
- [Background] Sause W, Kolesar P, Taylor S IV, Johnson D, Livingston R, Komaki R, Emami B, Curran W Jr, Byhardt R, Dar AR, Turrisi A 3rd. Final results of phase III trial in regionally advanced unresectable non-small cell lung cancer: Radiation Therapy Oncology Group, Eastern Cooperative Oncology Group, and Southwest Oncology Group. Chest. 2000 Feb;117(2):358-64. doi: 10.1378/chest.117.2.358. PMID 10669675
- [Background] Curran WJ, Scott C, Langer C, et al. Phase III comparision of sequential vs concurrent chemoradiation therapy for patients with unresectable stage III non-small cell lung cancer: initial report of RTOG 9410. Proc Am Soc Clin Oncol, 2000, 19: 484a.
- [Background] Furuse K, Fukuoka M, Kawahara M, Nishikawa H, Takada Y, Kudoh S, Katagami N, Ariyoshi Y. Phase III study of concurrent versus sequential thoracic radiotherapy in combination with mitomycin, vindesine, and cisplatin in unresectable stage III non-small-cell lung cancer. J Clin Oncol. 1999 Sep;17(9):2692-9. doi: 10.1200/JCO.1999.17.9.2692. PMID 10561343
- [Background] Auperin A, Le Pechoux C, Rolland E, Curran WJ, Furuse K, Fournel P, Belderbos J, Clamon G, Ulutin HC, Paulus R, Yamanaka T, Bozonnat MC, Uitterhoeve A, Wang X, Stewart L, Arriagada R, Burdett S, Pignon JP. Meta-analysis of concomitant versus sequential radiochemotherapy in locally advanced non-small-cell lung cancer. J Clin Oncol. 2010 May 1;28(13):2181-90. doi: 10.1200/JCO.2009.26.2543. Epub 2010 Mar 29. PMID 20351327
- [Background] Pfister DG, Johnson DH, Azzoli CG, Sause W, Smith TJ, Baker S Jr, Olak J, Stover D, Strawn JR, Turrisi AT, Somerfield MR; American Society of Clinical Oncology. American Society of Clinical Oncology treatment of unresectable non-small-cell lung cancer guideline: update 2003. J Clin Oncol. 2004 Jan 15;22(2):330-53. doi: 10.1200/JCO.2004.09.053. Epub 2003 Dec 22. No abstract available. PMID 14691125
- [Background] Strom HH, Bremnes RM, Sundstrom SH, Helbekkmo N, Flotten O, Aasebo U. Concurrent palliative chemoradiation leads to survival and quality of life benefits in poor prognosis stage III non-small-cell lung cancer: a randomised trial by the Norwegian Lung Cancer Study Group. Br J Cancer. 2013 Sep 17;109(6):1467-75. doi: 10.1038/bjc.2013.466. Epub 2013 Aug 20. PMID 23963145
- [Background] Strom HH, Bremnes RM, Sundstrom SH, Helbekkmo N, Aasebo U. Poor prognosis patients with inoperable locally advanced NSCLC and large tumors benefit from palliative chemoradiotherapy: a subset analysis from a randomized clinical phase III trial. J Thorac Oncol. 2014 Jun;9(6):825-33. doi: 10.1097/JTO.0000000000000184. PMID 24807158
- [Background] Lau DH, Crowley JJ, Gandara DR, Hazuka MB, Albain KS, Leigh B, Fletcher WS, Lanier KS, Keiser WL, Livingston RB. Southwest Oncology Group phase II trial of concurrent carboplatin, etoposide, and radiation for poor-risk stage III non-small-cell lung cancer. J Clin Oncol. 1998 Sep;16(9):3078-81. doi: 10.1200/JCO.1998.16.9.3078. PMID 9738578
- [Background] Davies AM, Chansky K, Lau DH, Leigh BR, Gaspar LE, Weiss GR, Wozniak AJ, Crowley JJ, Gandara DR; SWOG S9712. Phase II study of consolidation paclitaxel after concurrent chemoradiation in poor-risk stage III non-small-cell lung cancer: SWOG S9712. J Clin Oncol. 2006 Nov 20;24(33):5242-6. doi: 10.1200/JCO.2006.07.0268. PMID 17114656
- [Background] Robnett TJ, Machtay M, Vines EF, McKenna MG, Algazy KM, McKenna WG. Factors predicting severe radiation pneumonitis in patients receiving definitive chemoradiation for lung cancer. Int J Radiat Oncol Biol Phys. 2000 Aug 1;48(1):89-94. doi: 10.1016/s0360-3016(00)00648-9. PMID 10924976
- [Background] Torre-Bouscoulet L, Munoz-Montano WR, Martinez-Briseno D, Lozano-Ruiz FJ, Fernandez-Plata R, Beck-Magana JA, Garcia-Sancho C, Guzman-Barragan A, Vergara E, Blake-Cerda M, Gochicoa-Rangel L, Maldonado F, Arroyo-Hernandez M, Arrieta O. Abnormal pulmonary function tests predict the development of radiation-induced pneumonitis in advanced non-small cell lung Cancer. Respir Res. 2018 Apr 24;19(1):72. doi: 10.1186/s12931-018-0775-2. PMID 29690880
- [Background] Wang D, Zhu J, Sun J, Li B, Wang Z, Wei L, Yin Y, Sun H, Fu Z, Zhang X, Huo Z. Functional and biologic metrics for predicting radiation pneumonitis in locally advanced non-small cell lung cancer patients treated with chemoradiotherapy. Clin Transl Oncol. 2012 Dec;14(12):943-52. doi: 10.1007/s12094-012-0890-3. Epub 2012 Jul 20. PMID 22855174
- [Background] Dehing-Oberije C, De Ruysscher D, van Baardwijk A, Yu S, Rao B, Lambin P. The importance of patient characteristics for the prediction of radiation-induced lung toxicity. Radiother Oncol. 2009 Jun;91(3):421-6. doi: 10.1016/j.radonc.2008.12.002. Epub 2009 Jan 13. PMID 19147245
- [Background] Chen S, Zhou S, Zhang J, Yin FF, Marks LB, Das SK. A neural network model to predict lung radiation-induced pneumonitis. Med Phys. 2007 Sep;34(9):3420-7. doi: 10.1118/1.2759601. PMID 17926943
- [Background] Kong FM, Wang S. Nondosimetric risk factors for radiation-induced lung toxicity. Semin Radiat Oncol. 2015 Apr;25(2):100-9. doi: 10.1016/j.semradonc.2014.12.003. Epub 2014 Dec 15. PMID 25771414
- [Background] Inoue A, Kunitoh H, Sekine I, Sumi M, Tokuuye K, Saijo N. Radiation pneumonitis in lung cancer patients: a retrospective study of risk factors and the long-term prognosis. Int J Radiat Oncol Biol Phys. 2001 Mar 1;49(3):649-55. doi: 10.1016/s0360-3016(00)00783-5. PMID 11172945
- [Background] Ferrero C, Badellino S, Filippi AR, Focaraccio L, Giaj Levra M, Levis M, Moretto F, Torchio R, Ricardi U, Novello S. Pulmonary function and quality of life after VMAT-based stereotactic ablative radiotherapy for early stage inoperable NSCLC: a prospective study. Lung Cancer. 2015 Sep;89(3):350-6. doi: 10.1016/j.lungcan.2015.06.019. Epub 2015 Jun 26. PMID 26164208
- [Background] Blackstock AW, Socinski MA, Bogart J, et al; Cancer and Leukemia Group B. Induction plus concurrent chemotherapy with high-dose (74 Gy) 3-dimensional (3-D) thoracic radiotherapy in stage III non-small cell lung cancer. Preliminary report of Cancer and Leukemia Group B (CALGB) 30105. Proc Am Soc Clin Oncol 2006;24(18S):Abstr 7042.
- [Background] Lee CB, Socinski A, Lin L, et al. High-dose 3D chemoradiotherapy in stage III non-small cell lung cancer (NSCLC) at the University of North Carolina: long-term follow up and late complications. Proc Am Soc Clin Oncol 2006;24(18S):Abstr 7145
- [Background] Kong FM, Ten Haken RK, Schipper MJ, Sullivan MA, Chen M, Lopez C, Kalemkerian GP, Hayman JA. High-dose radiation improved local tumor control and overall survival in patients with inoperable/unresectable non-small-cell lung cancer: long-term results of a radiation dose escalation study. Int J Radiat Oncol Biol Phys. 2005 Oct 1;63(2):324-33. doi: 10.1016/j.ijrobp.2005.02.010. PMID 16168827
- [Background] Schild SE, McGinnis WL, Graham D, Hillman S, Fitch TR, Northfelt D, Garces YI, Shahidi H, Tschetter LK, Schaefer PL, Adjei A, Jett J. Results of a Phase I trial of concurrent chemotherapy and escalating doses of radiation for unresectable non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2006 Jul 15;65(4):1106-11. doi: 10.1016/j.ijrobp.2006.02.046. Epub 2006 May 26. PMID 16730134
- [Background] Bradley JD, Paulus R, Komaki R, Masters G, Blumenschein G, Schild S, Bogart J, Hu C, Forster K, Magliocco A, Kavadi V, Garces YI, Narayan S, Iyengar P, Robinson C, Wynn RB, Koprowski C, Meng J, Beitler J, Gaur R, Curran W Jr, Choy H. Standard-dose versus high-dose conformal radiotherapy with concurrent and consolidation carboplatin plus paclitaxel with or without cetuximab for patients with stage IIIA or IIIB non-small-cell lung cancer (RTOG 0617): a randomised, two-by-two factorial phase 3 study. Lancet Oncol. 2015 Feb;16(2):187-99. doi: 10.1016/S1470-2045(14)71207-0. Epub 2015 Jan 16. PMID 25601342
- [Background] Hanna N, Neubauer M, Yiannoutsos C, McGarry R, Arseneau J, Ansari R, Reynolds C, Govindan R, Melnyk A, Fisher W, Richards D, Bruetman D, Anderson T, Chowhan N, Nattam S, Mantravadi P, Johnson C, Breen T, White A, Einhorn L; Hoosier Oncology Group; US Oncology. Phase III study of cisplatin, etoposide, and concurrent chest radiation with or without consolidation docetaxel in patients with inoperable stage III non-small-cell lung cancer: the Hoosier Oncology Group and U.S. Oncology. J Clin Oncol. 2008 Dec 10;26(35):5755-60. doi: 10.1200/JCO.2008.17.7840. Epub 2008 Nov 10. PMID 19001323
- [Background] Spoelstra FO, Pantarotto JR, van Sornsen de Koste JR, Slotman BJ, Senan S. Role of adaptive radiotherapy during concomitant chemoradiotherapy for lung cancer: analysis of data from a prospective clinical trial. Int J Radiat Oncol Biol Phys. 2009 Nov 15;75(4):1092-7. doi: 10.1016/j.ijrobp.2008.12.027. Epub 2009 Mar 26. PMID 19327915
- [Background] Gielda BT, Marsh JC, Zusag TW, Faber LP, Liptay M, Basu S, Warren WH, Fidler MJ, Batus M, Abrams RA, Bonomi P. Split-course chemoradiotherapy for locally advanced non-small cell lung cancer: a single-institution experience of 144 patients. J Thorac Oncol. 2011 Jun;6(6):1079-86. doi: 10.1097/JTO.0b013e3182199a7c. PMID 21532501
- [Background] Belani CP, Choy H, Bonomi P, Scott C, Travis P, Haluschak J, Curran WJ Jr. Combined chemoradiotherapy regimens of paclitaxel and carboplatin for locally advanced non-small-cell lung cancer: a randomized phase II locally advanced multi-modality protocol. J Clin Oncol. 2005 Sep 1;23(25):5883-91. doi: 10.1200/JCO.2005.55.405. Epub 2005 Aug 8. PMID 16087941
- [Background] Curran W, Scott C, Langer C, et al. Phase III comparison of sequential vs concurrent chemoradiotherapy for patients (pts) with unresected stage III non-small cell lung cancer (NSCLC): report of Radiation Therapy Oncology Group (RTOG) 9410. Proc Am Soc Clin Oncol 2003;22:Abstr 2499.
- [Background] Albain KS, Swann RS, Rusch VW, Turrisi AT 3rd, Shepherd FA, Smith C, Chen Y, Livingston RB, Feins RH, Gandara DR, Fry WA, Darling G, Johnson DH, Green MR, Miller RC, Ley J, Sause WT, Cox JD. Radiotherapy plus chemotherapy with or without surgical resection for stage III non-small-cell lung cancer: a phase III randomised controlled trial. Lancet. 2009 Aug 1;374(9687):379-86. doi: 10.1016/S0140-6736(09)60737-6. Epub 2009 Jul 24. PMID 19632716
- [Background] Vokes EE, Herndon JE 2nd, Kelley MJ, Cicchetti MG, Ramnath N, Neill H, Atkins JN, Watson DM, Akerley W, Green MR; Cancer and Leukemia Group B. Induction chemotherapy followed by chemoradiotherapy compared with chemoradiotherapy alone for regionally advanced unresectable stage III Non-small-cell lung cancer: Cancer and Leukemia Group B. J Clin Oncol. 2007 May 1;25(13):1698-704. doi: 10.1200/JCO.2006.07.3569. Epub 2007 Apr 2. PMID 17404369
- [Background] Segawa Y, Kiura K, Takigawa N, Kamei H, Harita S, Hiraki S, Watanabe Y, Sugimoto K, Shibayama T, Yonei T, Ueoka H, Takemoto M, Kanazawa S, Takata I, Nogami N, Hotta K, Hiraki A, Tabata M, Matsuo K, Tanimoto M. Phase III trial comparing docetaxel and cisplatin combination chemotherapy with mitomycin, vindesine, and cisplatin combination chemotherapy with concurrent thoracic radiotherapy in locally advanced non-small-cell lung cancer: OLCSG 0007. J Clin Oncol. 2010 Jul 10;28(20):3299-306. doi: 10.1200/JCO.2009.24.7577. Epub 2010 Jun 7. PMID 20530281
- [Background] Fu KK, Pajak TF, Trotti A, Jones CU, Spencer SA, Phillips TL, Garden AS, Ridge JA, Cooper JS, Ang KK. A Radiation Therapy Oncology Group (RTOG) phase III randomized study to compare hyperfractionation and two variants of accelerated fractionation to standard fractionation radiotherapy for head and neck squamous cell carcinomas: first report of RTOG 9003. Int J Radiat Oncol Biol Phys. 2000 Aug 1;48(1):7-16. doi: 10.1016/s0360-3016(00)00663-5. PMID 10924966
- [Background] Saunders M, Dische S, Barrett A, Harvey A, Griffiths G, Palmar M. Continuous, hyperfractionated, accelerated radiotherapy (CHART) versus conventional radiotherapy in non-small cell lung cancer: mature data from the randomised multicentre trial. CHART Steering committee. Radiother Oncol. 1999 Aug;52(2):137-48. doi: 10.1016/s0167-8140(99)00087-0. PMID 10577699
- [Background] Petereit DG, Sarkaria JN, Chappell R, Fowler JF, Hartmann TJ, Kinsella TJ, Stitt JA, Thomadsen BR, Buchler DA. The adverse effect of treatment prolongation in cervical carcinoma. Int J Radiat Oncol Biol Phys. 1995 Jul 30;32(5):1301-7. doi: 10.1016/0360-3016(94)00635-X. PMID 7635769
- [Background] Begg AC, Hofland I, Van Glabekke M, et al. Predictive value of potential doubling time for radiotherapy of head and neck tumor patients: results from the EORTC cooperative trial 22851. Semin Radiat Oncol 1992;2:22-25.
- [Background] Desai N, Trieu V, Damascelli B, Soon-Shiong P. SPARC Expression Correlates with Tumor Response to Albumin-Bound Paclitaxel in Head and Neck Cancer Patients. Transl Oncol. 2009 May;2(2):59-64. doi: 10.1593/tlo.09109. PMID 19412420
- [Background] Desai N, Trieu V, Yao Z, Louie L, Ci S, Yang A, Tao C, De T, Beals B, Dykes D, Noker P, Yao R, Labao E, Hawkins M, Soon-Shiong P. Increased antitumor activity, intratumor paclitaxel concentrations, and endothelial cell transport of cremophor-free, albumin-bound paclitaxel, ABI-007, compared with cremophor-based paclitaxel. Clin Cancer Res. 2006 Feb 15;12(4):1317-24. doi: 10.1158/1078-0432.CCR-05-1634. PMID 16489089
- [Background] Green MR, Manikhas GM, Orlov S, Afanasyev B, Makhson AM, Bhar P, Hawkins MJ. Abraxane, a novel Cremophor-free, albumin-bound particle form of paclitaxel for the treatment of advanced non-small-cell lung cancer. Ann Oncol. 2006 Aug;17(8):1263-8. doi: 10.1093/annonc/mdl104. Epub 2006 Jun 1. PMID 16740598
- [Background] Rizvi NA, Riely GJ, Azzoli CG, Miller VA, Ng KK, Fiore J, Chia G, Brower M, Heelan R, Hawkins MJ, Kris MG. Phase I/II trial of weekly intravenous 130-nm albumin-bound paclitaxel as initial chemotherapy in patients with stage IV non-small-cell lung cancer. J Clin Oncol. 2008 Feb 1;26(4):639-43. doi: 10.1200/JCO.2007.10.8605. PMID 18235124
- [Background] Reynolds C, Barrera D, Jotte R, Spira AI, Weissman C, Boehm KA, Pritchard S, Asmar L. Phase II trial of nanoparticle albumin-bound paclitaxel, carboplatin, and bevacizumab in first-line patients with advanced nonsquamous non-small cell lung cancer. J Thorac Oncol. 2009 Dec;4(12):1537-43. doi: 10.1097/JTO.0b013e3181c0a2f4. PMID 19887966
- [Background] Socinski MA, Bondarenko I, Karaseva NA, Makhson AM, Vynnychenko I, Okamoto I, Hon JK, Hirsh V, Bhar P, Zhang H, Iglesias JL, Renschler MF. Weekly nab-paclitaxel in combination with carboplatin versus solvent-based paclitaxel plus carboplatin as first-line therapy in patients with advanced non-small-cell lung cancer: final results of a phase III trial. J Clin Oncol. 2012 Jun 10;30(17):2055-62. doi: 10.1200/JCO.2011.39.5848. Epub 2012 Apr 30. PMID 22547591
- [Background] Socinski MA, Okamoto I, Hon JK, Hirsh V, Dakhil SR, Page RD, Orsini J, Yamamoto N, Zhang H, Renschler MF. Safety and efficacy analysis by histology of weekly nab-paclitaxel in combination with carboplatin as first-line therapy in patients with advanced non-small-cell lung cancer. Ann Oncol. 2013 Sep;24(9):2390-6. doi: 10.1093/annonc/mdt235. Epub 2013 Jul 10. PMID 23842283
- [Background] Hasegawa T, Futamura Y, Horiba A, Yoshida T, Suzuki T, Kato T, Kaito D, Ohno Y, Iida T, Hayashi S, Sawa T. A phase II study of nab-paclitaxel plus carboplatin in combination with thoracic radiation in patients with locally advanced non-small-cell lung cancer. J Radiat Res. 2016 Jan;57(1):50-4. doi: 10.1093/jrr/rrv062. Epub 2015 Oct 5. PMID 26442970
- [Background] Lammers PE, Lu B, Horn L, Shyr Y, Keedy V. nab-Paclitaxel in Combination With Weekly Carboplatin With Concurrent Radiotherapy in Stage III Non-Small Cell Lung Cancer. Oncologist. 2015 May;20(5):491-2. doi: 10.1634/theoncologist.2015-0030. Epub 2015 Apr 6. PMID 25845992
- [Background] Kaira K, Tomizawa Y, Imai H, Sakurai R, Matsuura M, Yoshii A, Ochiai M, Kotake M, Ebara T, Saitoh JI, Sunaga N, Minato K, Saito R, Hisada T. Phase I study of nab-paclitaxel plus carboplatin and concurrent thoracic radiotherapy in patients with locally advanced non-small cell lung cancer. Cancer Chemother Pharmacol. 2017 Jan;79(1):165-171. doi: 10.1007/s00280-016-3217-1. Epub 2016 Dec 19. PMID 27995307
- [Background] Kawano Y, Sasaki T, Yamaguchi H, Hirano K, Horiike A, Satouchi M, Hosokawa S, Morinaga R, Komiya K, Inoue K, Fujita Y, Toyozawa R, Kimura T, Takahashi K, Nishikawa K, Kishimoto J, Nakanishi Y, Okamoto I. Phase I/II study of carboplatin plus nab-paclitaxel and concurrent radiotherapy for patients with locally advanced non-small cell lung cancer. Lung Cancer. 2018 Nov;125:136-141. doi: 10.1016/j.lungcan.2018.09.014. Epub 2018 Sep 18. PMID 30429011